CLINICAL TRIAL: NCT03491865
Title: Peer-to-peer Social Media Diffusion of Tobacco and ENDS Use Prevention Messages
Brief Title: Peer-to-peer Tobacco and ENDS Prevention
Acronym: PPSM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: unfunded
Sponsor: Real Prevention, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 284105
Record Dates: First submitted 2018-04-02; First posted 2018-04-09 (Actual); Last update posted 2019-09-11 (Actual); Status verified 2019-09

CONDITIONS: Substance Use
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- REAL media Plus (Experimental): Participants in this group will be assigned to use the REAL media Plus curriculum.
  Interventions: Behavioral: REAL media Plus curriculum
- programming as usual (No Intervention): Participants in this group will participate in their usual school curriculum. They will have the opportunity to use the REAL media Plus curriculum at the conclusion of the study.

INTERVENTIONS:
Behavioral: REAL media Plus curriculum — REAL media Plus is a 7-level, interactive, self-paced, e-learning media literacy curriculum to prevent youth smoking and vaping use.
  Arms: REAL media Plus

SUMMARY:
In Phase I, the REAL media Plus prototype will be developed and a usability test conducted among students and teachers.

In Phase II a group randomized trial will be conducted among 27 high schools to evaluate the effects of REAL media Plus on smoking and vaping.

DETAILED DESCRIPTION:
In Phase I, participants will participate in pilot and usability tests of the curriculum prototype. For the pilot test, teachers and students will use the curriculum prototype and then be interviewed about it. For the usability test, students and teachers will use the revised curriculum and be interviewed/complete short survey. Teachers will provide consent and students will have parental consent and their own assent.

In Phase II, a group randomized trial will be conducted during Spring semester 2020 among 9th grade student in 27 high schools in the Hillsborough County Public School system randomly assigned to treatment and control (14 treatment and 13 control). All students will complete a pretest survey. Students in two health classes in treatments schools will participate in the REAL media Plus curriculum and complete a short immediate posttest survey to rate their experience. All students will then complete two posttests. Students will have parental consent and provide their own assent.

ELIGIBILITY:
Inclusion Criteria:

Attendance at participating schools; 9th grade student status (for student participants, both phase 1 and 2); status as a teacher/counselor (for phase 1); written parental consent and assent from students (phase 1 and 2); written consent from counselors/teachers (phase 1); and all individuals must be willing to participate.

Exclusion Criteria:

Exclusion criteria include the inability to speak or read American English, use a computer, or navigate the Internet and, for youth, lack of parental consent.

Ages: 13 Years to 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2018-09-01 (Estimated); Primary Completion 2021-05-31 (Estimated); Study Completion 2021-05-31 (Estimated)

PRIMARY OUTCOMES:
Smoking and Vaping Use | Change in llifetime (e.g., ever tried) use from baseline to 9 months post baseline
  Change in 5-item Lifetime Substance Use Measure Self reported lifetime use of (e.g., whether you ever tried) cigarettes and vaping. Response options include Yes and No.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hecht, PhD, Principal Investigator — Real Prevention, LLC
Locations (1):
- REAL Prevention LLC, Clifton, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided